CLINICAL TRIAL: NCT02248233
Title: Nimodipine for Treating Acute Massive Cerebral Infarction: a Randomized, Double-blind, Controlled Clinical Study
Brief Title: Nimodipine for Treating Acute Massive Cerebral Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fengtian Hospital (Other)
Responsible Party: Principal Investigator, Runhui Li, Director, Fengtian Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FengtianH-RHL-001
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Cerebral Infarction
Keywords: nimodipine; acute massive cerebral infarction; Cerebral Infarction; optimal therapeutic time window; optimal dose; multi-center
MeSH Terms: conditions — Cerebral Infarction | interventions — Nimodipine; Sodium Chloride; Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline + citicoline (Experimental): The control group will receive physiological saline + citicoline 2.0 g, once a day, via intravenous drip, for 10 consecutive days. Patients will receive additional drugs to treat dehydration, prevent infection and upper gastrointestinal bleeding, and maintain water and electrolyte balance. Patients with complications will receive symptomatic treatment.
  Interventions: Drug: Saline + citicoline
- Nimodipine (Experimental): The treatment group will receive 10 mg of nimodipine in 500 ml of physiological saline via intravenous drip, at a rate of 1-2 drops per minute initially, increasing gradually until systolic pressure decreases by 10 mmHg. Maximum drip speed is 10 drops/minute, administered once a day for 7 consecutive days. The nimodipine must be kept in the dark. Blood pressure and heart rate will be monitored throughout the administration period.
  Patients in control group will receive additional drugs to treat dehydration, prevent infection and upper gastrointestinal bleeding, and maintain water and electrolyte balance. Patients with complications will receive symptomatic treatment.
  Interventions: Drug: Nimodipine

INTERVENTIONS:
Drug: Nimodipine — Jiangsu Jichuan Pharmaceutical Co., Ltd., Jiangsu Province, China
  Other Names: The treatment group
  Arms: Nimodipine
Drug: Saline + citicoline — physiological saline + citicoline 2.0 g, once a day, via intravenous drip, for 10 consecutive days.
  Other Names: The control group
  Arms: Saline + citicoline

SUMMARY:
Massive cerebral infarction is an ischemic stroke caused by complete blockage of the internal carotid artery, middle cerebral artery, or their cortical branches. The widespread infarction, pathological severity and high fatality rate associated with massive cerebral infarction pose a major threat to affected patients. However, there is a lack of unified diagnostic criteria. Many researchers use Adams' classification, in which massive cerebral infarction is diagnosed when the following criteria are met: infarct size > 13 cm2; a major brain-feeding artery is involved; the focal site affects more than two cerebral lobes; infarct diameter line ≥ 3 cm in internal capsule of striatum.

Prolonged cerebral ischemia/reperfusion can induce complex secondary changes in brain tissue, so the use of neuroprotective agents is very important. Remarkable progress has been made over the last decade in understanding the protective effect of calcium antagonists against cerebral ischemia. In particular, the liposoluble dihydropyridine Ca2+ antagonist nimodipine selectively acts on cerebral vessels and neurons and can protect ischemic brain tissue, providing a new way of treating ischemic cerebrovascular disease.

Preclinical and clinical tests have shown that nimodipine has a protective effect on ischemic brain tissue, and indicate that patients should take the drug as soon as possible. However, there are no reports of double-blind, randomized, controlled clinical trials addressing the administration of nimodipine via intravenous drip within the time window for successful treatment of acute massive cerebral infarction.

DETAILED DESCRIPTION:
In the clinic, physicians are reluctant to use thrombolysis, Defibrase and anticoagulation therapy because of the severity of symptoms, poor prognosis, risk of hemorrhage and high fatality rate that occur with acute massive cerebral infarction. Nimodipine, as a selective Ca2+ antagonist, is highly liposoluble, effectively crosses the blood-brain barrier, selectively acts on intracranial blood vessels, and is an accepted neuroprotective agent that can be applied in the clinic. The aim of the present study is to perform a double-blind, randomized and controlled trial of the clinical efficacy and safety of nimodipine administered as an intravenous drip in the early stages of acute massive cerebral infarction.

Patients will receive nimodipine within 3 days of infarction onset. We will closely monitor the following: (1) Blood pressure and heart rate of the patient before treatment, since nimodipine is contraindicated in patients with hypotension and low heart rate. Where blood pressure is ≥ 100/80 mmHg and heart rate ≥ 60 BPM, nimodipine will be administered. (2) Speed of infusion. This should not be too fast; we suggest 1-2 drops per minute initially, increasing gradually until the drop in systolic pressure exceeds 10 mmHg. The average drip speed should be 6-8 drops/minute, and the fastest drip speed 10 drops/minute. (3) During the infusion, physicians should monitor adverse reactions such as headache, dizziness, flushing or sweating. If any occur, the infusion speed must be reduced. If the patients remain uncomfortable, nimodipine should be withdrawn. (4) Liver and kidney function should be monitored throughout nimodipine administration.

Although nimodipine is relatively safe, there is still a risk of some adverse effects, such as cardiovascular system reactions (blood pressure decreases, bradycardia, angina, and atrioventricular block), headache, dizziness, edema, and liver and kidney dysfunction. It is necessary to determine the optimal therapeutic time window and dose of nimodipine in multi-center, large-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* First onset at age ≤ 80 years, no other severe medical complications;
* Clear consciousness or mild disturbance of consciousness; paralysis of upper and lower extremities on one side with grade 0-3 muscle strength in paralyzed limbs;
* CT reveals early massive cerebral infarction (without cerebral hemorrhage or old infarction);
* Blood pressure within, or higher than, the normal range.

Exclusion Criteria:

* Clinical manifestations are noticeably improved before treatment;
* Disorders of consciousness, manifesting as severe lethargy or coma;
* Mild neurological deficits, such as pure sensory disturbances, ataxia, dysarthria, and hemiparesis;
* Severe hypotension (systolic pressure < 90 mmHg, diastolic pressure < 60 mmHg);
* Heart rate < 60 BPM; sinus bradycardia;
* Severe heart, brain or kidney dysfunction, or malignant tumor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Neurological deficits | up to 90 days
  Neurological deficits after stroke will be assessed using the National Institute of Health Stroke Scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Runhui Li, M.D., Principal Investigator — Central Hospital Affiliated to Shenyang Medical Collage